CLINICAL TRIAL: NCT01086124
Title: Objective Systolic Function Recuperation Assessed by Echocardiography
Acronym: ROSE
Status: Completed | Type: Observational
Sponsor: Paul Farand (Other)
Responsible Party: Sponsor-Investigator, Paul Farand, MD, Université de Sherbrooke
Organization: Université de Sherbrooke (Other)
Other Study IDs: 10-010
Record Dates: First submitted 2010-03-11; First posted 2010-03-12 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-07

CONDITIONS: Myocardial Infarction; Left Ventricular Systolic Dysfunction; Anterior Akinesis; Apical Akinesis
Keywords: echocardiography; ST elevation myocardial infarction; Heart failure; Coronary artery disease; Cardiovascular diseases
MeSH Terms: conditions — Myocardial Infarction; Ventricular Dysfunction, Left; ST Elevation Myocardial Infarction; Heart Failure; Coronary Artery Disease; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Echocardiography 1 month: Patients will all have an echocardiography 1 month post myocardial infarction and 3 months post myocardial infarction

SUMMARY:
The purpose of this study is to evaluate left ventricular systolic ejection fraction and anterior or apical akinesis 1 month and 3 months after a myocardial infarction treated with primary PCI to determine whether improvement at 1 month differs from improvement at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years old
* ST elevation myocardial infarction treated with primary PCI
* Anterior or apical akinesis and left ventricular ejection fraction ≤ 45% on early echocardiography (48hours - 7 days post myocardial infarction)
* Initial ECG showing at least 1 mm ST elevation in 2 leads corresponding to the same vascular territory

Exclusion Criteria:

* Known left ventricular systolic dysfunction before myocardial infarction
* Left bundle branch block
* Vital prognosis less than 6 months
* Cardiogenic shock
* Rescue PCI
* Sub-optimal echocardiographic imaging (contrast use is allowed)
* Significant valvular heart disease (moderate or severe)
* Surgical revascularization
* Pregnancy or breastfeeding
* Incapacity to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to teaching hospital or sent from community hopitals to teaching hospital for primary PCI
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2010-03; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Left ventricular ejection fraction recuperation 1 month post myocardial infarction | 1 month post myocardial infarction
  Left ventricular ejection fraction recuperation 1 month post myocardial infarction as compared with the left ejection fraction 3 months post myocardial infarction

SECONDARY OUTCOMES:
Anterior and apical akinesis recuperation 1 month post myocardial infarction | 1 month post myocardial infarction
  Anterior and apical akinesis recuperation 1 month post myocardial infarction as compared with 3 months post myocardial infarction

CONTACTS AND LOCATIONS:
Overall Officials: Paul Farand, md, Principal Investigator — Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Locations (1):
- Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec, Canada